CLINICAL TRIAL: NCT03116542
Title: A Study of 18F-FLT Positron Emission Tomography/Computed Tomography (PET/CT) Imaging in Cases of Prefibrotic/Early Primary Myelofibrosis (PMF) and Essential Thrombocythemia (ET)
Brief Title: 18F-FLT (PET/CT) in Prefibrotic/Early Primary Myelofibrosis and Essential Thrombocythemia
Acronym: PMF/ET-FLT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16287/16
Record Dates: First submitted 2017-04-04; First posted 2017-04-17 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2019-11

CONDITIONS: Essential Thrombocythemia; Primary Myelofibrosis, Fibrotic Stage; Primary Myelofibrosis, Prefibrotic Stage
MeSH Terms: conditions — Thrombocythemia, Essential; Primary Myelofibrosis | interventions — Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Diagnostic (18F-FLT PET/CT) (Experimental): Patients undergo 18F-FLT (3'-18Fluoro-3'-deoxy-L-thymidine) PET/CT (Positron Emission Tomography/Computed Tomography) at baseline. No specific dietary restrictions or hydration are required for FLT-PET scans, however, patients will be urged to drink plenty of water before and after the PET studies. [18F] FLT will be prepared by the cyclotron core facility and assessed for quality control following "good manufacturing practice" criteria. The radiopharmaceutical will immediately be brought to the Molecular Imaging and Therapy Service Radiopharmacy for dispensation in the PET suite. For each scan, patients will receive approximately up to 370 MBq (target of 10 mCi) [18F] FLT by intravenous infusion.
  Interventions: Device: Diagnostic (18F-FLT PET/CT)

INTERVENTIONS:
Device: Diagnostic (18F-FLT PET/CT) — The tracer compound [F-18] FLT will be injected into the patient's veins in a small volume of normal saline solution. The PET scan data collection is started immediately and is continued for 2 hours.
  Other Names: 18F-FLT PET/CT; 3'-Deoxy-3'-(18F) Fluorothymidine; 3'-deoxy-3'-[18F]fluorothymidine; Fluorothymidine F 18

SUMMARY:
The main purpose of this project is to study the uptake pattern of FLT-PET in cases, and it is value in assessing the malignant hematopoiesis in cases of Pre-PMF and ET, regarding diagnosis, staging and monitoring response to therapy. Identifying different patterns of uptake in patients with Pre-PMF and ET in various clinical settings.

Evaluating FLT-PET as a novel non-invasive technique in cases with Pre-PMF and ET, in comparison to the standard bone marrow biopsy about disease diagnosis, assessment of disease activity, detection of transformation, monitoring of treatment response and grading of fibrosis.Study the ability of FLT-PET to differentiate between Pre-PMF and ET.

the investigators also aim to examine the association of FLT-PET uptake patterns with different genetic makeup (JAK2 (Janus kinase 2), CALR (Calreticulin), MPL (myeloproliferative leukemia protein), or Triple negative disease) or allele burden in cases of Pre-PMF and ET.

DETAILED DESCRIPTION:
PET with fluorodeoxy glucose combined with computed tomography is a major tool for the diagnosis, staging, and monitoring of treatment response in clinical oncology. 3'-18Fluoro-3'-deoxy-L-thymidine (18F-FLT) is a PET radiotracer that quickly accumulates in proliferating cells and can be used to assess tumor cell proliferation in various cancers as PET radiotracer offers a non-invasive assessment of cell proliferation in vivo.

Myeloproliferative Neoplasms (MPNs) are clonal hematopoietic stem disorders characterized by high rate of effective proliferation of one or more cell lineage. MPNs are overlapping syndromes that can progress to fibrotic stage or evolute into acute leukemia. Preliminary results of a pilot study (5) suggested that this technique could be useful to assess bone marrow (BM) activity and extramedullary hematopoiesis in patients with Myelofibrosis (MF).

The current standard for follow- up of these patients is based on pathological markers (peripheral blood counts and/ bone marrow histomorphology) and molecular markers. Although, bone marrow examination could be considered as a standard gold method as it gives detailed information about cellularity, the morphology of each lineage, a degree of fibrosis, transformation and dysplastic features. However, many patients are reluctant to go for this invasive technique which precludes precise assessment of disease activity at the desirable frequencies. Non- invasive techniques which may act as the good clinical surrogate are lacking.

The objective of this study is to study the uptake pattern of FLT-PET in cases, and it is value in assessing the malignant hematopoiesis in cases of Pre-PMF and ET, regarding diagnosis, staging and monitoring response to therapy.

Identifying different patterns of uptake in patients with Pre-PMF and ET in various clinical settings.

Evaluating FLT-PET as a novel non-invasive technique in cases with Pre-PMF and ET, in comparison to the standard bone marrow biopsy about disease diagnosis, assessment of disease activity, detection of transformation, monitoring of treatment response and grading of fibrosis.

Study the ability of FLT-PET to differentiate between Pre-PMF and ET. the investigators also aim to investigate the association of FLT-PET uptake patterns with different genetic makeup (JAK2, CALR, MPL, or Triple negative disease) or allele burden in cases of Pre-PMF and ET.

ELIGIBILITY:
Inclusion Criteria:

Age 18 year old or above Patient accept to sign inform consent ECOG (Eastern Cooperative Oncology Group) performance less than or equal 2

* Cases fulfilling WHO (World Health Organization) 2016 diagnostic criteria for PMF:

WHO criteria for prefibrotic/early primary myelofibrosis (prePMF)

Major criteria:

1. Megakaryocytic proliferation and atypia, without reticulin fibrosis > grade 1*, accompanied by increased age-adjusted BM cellularity, granulocytic proliferation and often decreased erythropoiesis
2. Not meeting the WHO criteria for BCR-ABL1+ ((BCR-ABL = fusion gene from BCR (breakpoint cluster region gene/BCR gene product) and ABL (Abelson proto-oncogene)) CML (chronic myelogenous leukemia), PV (Polycythemia Vera), ET, myelodysplastic syndromes, or other myeloid neoplasms
3. Presence of JAK2, CALR or MPL mutation or in the absence of these mutations, presence of another clonal marker**or absence of minor reactive BM reticulin fibrosis.

Minor criteria:

Presence of at least one of the following, confirmed in two consecutive determinations:

1. Anemia not attributed to a comorbid condition
2. Leukocytosis >11 x 109/L
3. Palpable splenomegaly
4. LDH (Lactate dehydrogenase) increased to above upper normal limit of institutional reference range.

Diagnosis of prePMF requires meeting all three major criteria, and at least one minor criterion **in the absence of any of the 3 major clonal mutations, the search for the most frequent accompanying gene mutations (e.g. ASXL1, EZH2, TET2, IDH1/IDH2, SRSF2, SF3B1) are of help in determining the clonal nature of the disease.

*** minor (grade 1) reticulin fibrosis secondary to infection, autoimmune disorder or other chronic inflammatory conditions, hairy cell leukemia or other lymphoid neoplasm, metastatic malignancy, or toxic (chronic) myelopathies

WHO diagnostic criteria essential thrombocythemia Major criteria Platelet count ≥450 × 109/L Bone marrow biopsy showing proliferation mainly of the megakaryocyte lineage with increased numbers of enlarged, mature megakaryocytes with hyperlobulated nuclei. No significant increase or left shift in neutrophil granulopoiesis or erythropoiesis and very rarely minor (grade 1) increase in reticulin fibers.

Not meeting WHO criteria for BCR-ABL1+ CML, PV, PMF, myelodysplastic syndromes, or other myeloid neoplasms Presence of JAK2, CALR, or MPL mutation Minor criterion Presence of a clonal marker or absence of evidence for reactive thrombocytosis Diagnosis of ET requires meeting all 4 major criteria or the first 3 major criteria and the minor criterion

Exclusion Criteria:

* Patient not fulfilling the inclusion criteria.
* Vulnerable groups: pregnant, minors, prisoners will not be included.
* Bone marrow will be collected as part of the routine diagnostic work-up. No extra bone marrow material will be collected solely for the aim of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2017-05-07 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with 50% or more uptake of FLT-PET in patients with Prefibrotic/Early Primary Myelofibrosis (PMF) and Essential Thrombocythemia (ET) 12 months from the baseline | 12 Months
  Evaluate the uptake of 3'-deoxy-3'-[18F] fluorothymidine (FLT) positron emission tomography/computed tomography (PET) imaging and it is value in assessing the malignant hematopoiesis in patients with Prefibrotic/Early Primary Myelofibrosis (PMF) and Essential Thrombocythemia (ET).

SECONDARY OUTCOMES:
Reduction in at least 50% of the allele burden of different mutations (JAK-2, MPL, CALR) and its expression on FLT- PET uptake pattern 12 moths from the baseline | 12 Months
  Effect of different mutations (JAK-2, MPL, CALR) expression and allele burden on FLT- PET uptake pattern

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Cancer Care & Research (NCCCR), Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pikman Y, Lee BH, Mercher T, McDowell E, Ebert BL, Gozo M, Cuker A, Wernig G, Moore S, Galinsky I, DeAngelo DJ, Clark JJ, Lee SJ, Golub TR, Wadleigh M, Gilliland DG, Levine RL. MPLW515L is a novel somatic activating mutation in myelofibrosis with myeloid metaplasia. PLoS Med. 2006 Jul;3(7):e270. doi: 10.1371/journal.pmed.0030270. PMID 16834459
- [Background] Beer PA, Campbell PJ, Scott LM, Bench AJ, Erber WN, Bareford D, Wilkins BS, Reilly JT, Hasselbalch HC, Bowman R, Wheatley K, Buck G, Harrison CN, Green AR. MPL mutations in myeloproliferative disorders: analysis of the PT-1 cohort. Blood. 2008 Jul 1;112(1):141-9. doi: 10.1182/blood-2008-01-131664. Epub 2008 May 1. PMID 18451306
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254
- [Background] Agool A, Schot BW, Jager PL, Vellenga E. 18F-FLT PET in hematologic disorders: a novel technique to analyze the bone marrow compartment. J Nucl Med. 2006 Oct;47(10):1592-8. PMID 17015893
- [Background] Chalkidou A, Landau DB, Odell EW, Cornelius VR, O'Doherty MJ, Marsden PK. Correlation between Ki-67 immunohistochemistry and 18F-fluorothymidine uptake in patients with cancer: A systematic review and meta-analysis. Eur J Cancer. 2012 Dec;48(18):3499-513. doi: 10.1016/j.ejca.2012.05.001. Epub 2012 May 31. PMID 22658807
- [Background] Chen W, Cloughesy T, Kamdar N, Satyamurthy N, Bergsneider M, Liau L, Mischel P, Czernin J, Phelps ME, Silverman DH. Imaging proliferation in brain tumors with 18F-FLT PET: comparison with 18F-FDG. J Nucl Med. 2005 Jun;46(6):945-52. PMID 15937304
- [Background] Ott K, Herrmann K, Schuster T, Langer R, Becker K, Wieder HA, Wester HJ, Siewert JR, zum Buschenfelde CM, Buck AK, Wilhelm D, Ebert MP, Peschel C, Schwaiger M, Lordick F, Krause BJ. Molecular imaging of proliferation and glucose utilization: utility for monitoring response and prognosis after neoadjuvant therapy in locally advanced gastric cancer. Ann Surg Oncol. 2011 Nov;18(12):3316-23. doi: 10.1245/s10434-011-1743-y. Epub 2011 May 3. PMID 21537865
- [Background] Ott K, Rachakonda PS, Panzram B, Keller G, Lordick F, Becker K, Langer R, Buechler M, Hemminki K, Kumar R. DNA repair gene and MTHFR gene polymorphisms as prognostic markers in locally advanced adenocarcinoma of the esophagus or stomach treated with cisplatin and 5-fluorouracil-based neoadjuvant chemotherapy. Ann Surg Oncol. 2011 Sep;18(9):2688-98. doi: 10.1245/s10434-011-1601-y. Epub 2011 Feb 24. PMID 21347786
- [Background] Graf N, Herrmann K, den Hollander J, Fend F, Schuster T, Wester HJ, Senekowitsch-Schmidtke R, zum Buschenfelde CM, Peschel C, Schwaiger M, Dechow T, Buck AK. Imaging proliferation to monitor early response of lymphoma to cytotoxic treatment. Mol Imaging Biol. 2008 Nov-Dec;10(6):349-55. doi: 10.1007/s11307-008-0162-3. Epub 2008 Aug 14. PMID 18704591
- [Background] Leonard JP, LaCasce AS, Smith MR, Noy A, Chirieac LR, Rodig SJ, Yu JQ, Vallabhajosula S, Schoder H, English P, Neuberg DS, Martin P, Millenson MM, Ely SA, Courtney R, Shaik N, Wilner KD, Randolph S, Van den Abbeele AD, Chen-Kiang SY, Yap JT, Shapiro GI. Selective CDK4/6 inhibition with tumor responses by PD0332991 in patients with mantle cell lymphoma. Blood. 2012 May 17;119(20):4597-607. doi: 10.1182/blood-2011-10-388298. Epub 2012 Mar 1. PMID 22383795
- [Background] Zhang CC, Yan Z, Li W, Kuszpit K, Painter CL, Zhang Q, Lappin PB, Nichols T, Lira ME, Affolter T, Fahey NR, Cullinane C, Spilker M, Zasadny K, O'Brien P, Buckman D, Wong A, Christensen JG. [(18)F]FLT-PET imaging does not always "light up" proliferating tumor cells. Clin Cancer Res. 2012 Mar 1;18(5):1303-12. doi: 10.1158/1078-0432.CCR-11-1433. Epub 2011 Dec 14. PMID 22170262
- [Background] Shields AF, Grierson JR, Dohmen BM, Machulla HJ, Stayanoff JC, Lawhorn-Crews JM, Obradovich JE, Muzik O, Mangner TJ. Imaging proliferation in vivo with [F-18]FLT and positron emission tomography. Nat Med. 1998 Nov;4(11):1334-6. doi: 10.1038/3337. PMID 9809561
- [Background] Vesselle H, Salskov A, Turcotte E, Wiens L, Schmidt R, Jordan CD, Vallieres E, Wood DE. Relationship between non-small cell lung cancer FDG uptake at PET, tumor histology, and Ki-67 proliferation index. J Thorac Oncol. 2008 Sep;3(9):971-8. doi: 10.1097/JTO.0b013e31818307a7. PMID 18758298
- [Derived] Yassin MA, Nehmeh SA, Nashwan AJ, Kohla SA, Mohamed SF, Ismail OM, Sabbagh AA, Ibrahim F, Soliman DS, Szabados L, Fayad H. A study of 18F-FLT positron emission tomography/computed tomography imaging in cases of prefibrotic/early primary myelofibrosis and essential thrombocythemia. Medicine (Baltimore). 2020 Nov 6;99(45):e23088. doi: 10.1097/MD.0000000000023088. PMID 33157979